CLINICAL TRIAL: NCT05395247
Title: Evaluation gériatrique Avant Transplantation rénale
Brief Title: Geriatric Assessment for Older Kidney Transplantation Candidates
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Cédric VILLAIN, Principal investigator, University Hospital, Caen
Other Study IDs: 1154
Record Dates: First submitted 2022-02-08; First posted 2022-05-27 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; kidney transplantation; comprehensive geriatric assessment
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Geriatric assessment — Geriatric assessment by a trained nurse and a geriatrician for older kidney transplantation candidates in Caen University Hospital. The geriatric assessment includes a evaluation of cognitive functions, depressive symptoms, risk of fall, nutrition, frailty, and functional status.

SUMMARY:
Geriatric assessment is now widely used to decide whether older patients with chronic kidney disease should be put on the kidney transplantation waiting list. This study aims to evaluate the association between Geriatric assessment and inscription on kidney transplantation.

DETAILED DESCRIPTION:
There is a high proportion of older patients among patients with kidney failure, raising the question of the access to kidney transplantation within these patients. Geriatric assessment is now widely used to decide whether older patients with chronic kidney disease should be put on the kidney transplantation waiting list.

This study aims to evaluate the association between Geriatric assessment and inscription on kidney transplantation. Secondary objectives includes the analysis of the association between Geriatric assessment and:

* post-kidney transplantation outcomes
* quality of life.

It also includes the evolution of Geriatric assessment while still on waiting list and after kidney transplantation.

This study takes place in an University Hospital in Caen, France. This hospital is the only one performing kidney transplantation in the three French departments around. Candidates for kidney transplantation older than 70 years are systematically evaluated by a trained nurse and a geriatrician to perform a comprehensive geriatric assessment, evaluating cognitive functions, risk of fall, nutrition, frailty, functional status, and depressive symptoms. These patients are followed-up each year while still on the waiting list, and once after kidney transplantation. All patients evaluated within this consultation are proposed to enter the study. Patients are excluded in case of refusal or if they are unable to provide informed consent. The inclusion began in January 2019.

ELIGIBILITY:
Inclusion Criteria:

* All patients addressed for Geriatric assessment before inscription on kidney transplantation waiting list in Caen University Hospital, France

Exclusion Criteria:

* Patient refusal
* Patient unable to provide informed consent

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients with chronic kidney disease stages 4-5 treated or not by dialysis or kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Inscription on kidney transplantation waiting list | 6 months
  Inscription on kidney transplantation waiting list

SECONDARY OUTCOMES:
Length of hospitalization in the year following kidney transplantation | 1 year after kidney transplantation
  Units: days
Delayed renal recovery following kidney transplantation | 1 week after kidney transplantation
  Dialysis requirement during the first week after kidney transplantation
Mortality | 1 year after kidney transplantation
  Death in the year following kidney transplantation

OTHER OUTCOMES:
Evolution of quality of life while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Assessed by the SF12 score before and in the year after kidney transplantation
Evolution of cognitive functions while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Cognitive functions assessed by MMSE score
Evolution of executive functions while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Executive functions assessed by BREF test
Evolution of mood while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Mood assessed by the mini GDS scale
Evolution of frailty while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Frailty assessed by the Rockwood scale
Evolution of functionnal status while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Functionnal status assessed by activities of daily living scales
Evolution of functionnal status while on waiting list and after kidney transplantation | 1 year after kidney transplantation
  Functionnal status assessed by the walk speed in m/s

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Villain, MD, PhD, Principal Investigator — Department of Geriatrics, Caen University Hospital, Caen, France
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
Data would be available on reasonable request